CLINICAL TRIAL: NCT05099952
Title: Sleep and Circadian Rhythm Study in Head and Neck Cancer Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institute-no accruals
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: I 864421; NCI-2021-09748 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 864421 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2021-09-29; First posted 2021-10-29 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Counseling; Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm I - BBT-CI (Experimental): Patients participate in BBT-CI over 60 minutes for 2 sessions and phone calls over 15 minutes once weekly for 4 weeks.
  Interventions: Other: Educational Intervention; Other: Questionnaire Administration
- Arm II- therapist (Active Comparator): Patients meet with therapist over 60 minutes for 2 sessions and phone calls over 15 minutes once weekly for 4 weeks.
  Interventions: Other: Counseling; Other: Questionnaire Administration
- Observational Study (Experimental): Patients wear actigraphy watch and complete sleep log at baseline (over the weekend prior to first day of CRT), and weeks 1, 3, and 6 during treatment. Patients also undergo collection of cheek cell samples and may undergo collection of blood samples at weeks 1, 3 and 6 during treatment. Patients' medical records are also reviewed.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Other: Medical Device Usage and Evaluation; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of cheek cell and blood samples
  Other Names: Biological Sample Collection
  Arms: Observational Study
Other: Counseling — Meet with therapist
  Other Names: Counseling Intervention
  Arms: Arm II- therapist
Other: Educational Intervention — Participate in BBT-CI sessions
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm I - BBT-CI
Other: Electronic Health Record Review — Medical records are reviewed
  Arms: Observational Study
Other: Medical Device Usage and Evaluation — Wear actigraphy watch
  Arms: Observational Study
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies the effect and underlying mechanisms of sleep and circadian rhythm factors on oral mucositis pain in head and neck cancer patients treated by chemoradiotherapy. Poor sleep may have a correlation to increased pain. A behavioral intervention, Brief Behavioral Therapy for Cancer related Insomnia, may improve patients' sleep and may also reduce oral mucositis pain.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine the effect and underlying mechanisms of sleep and circadian rhythm factors on oral mucositis pain in head and neck cancer patients treated by chemoradiotherapy.

Ia. To assess the impact of chemo-radiotherapy (CRT) on the onset and duration of sleep disturbance in head and neck carcinoma (HNC) patients, and identify factors that trigger or aggravate sleep disturbance.

Ib. To examine the effect of the association between sleep and CRT-induced oral mucositis (OM) pain.

SECONDARY OBJECTIVE:

I. To examine the pathways by which sleep disturbance may aggravate radiation-induced OM pain.

OUTLINE:

OBSERVATIONAL STUDY: Patients wear actigraphy watch and complete sleep log at baseline (over the weekend prior to first day of CRT), and weeks 1, 3, and 6 during treatment. Patients also undergo collection of cheek cell samples and may undergo collection of blood samples at weeks 1, 3 and 6 during treatment. Patients' medical records are also reviewed.

INTERVENTION STUDY: Patients are randomized to 1 of 2 arms.

ARM I: Patients participate in BBT-CI over 60 minutes for 2 sessions and phone calls over 15 minutes once weekly for 4 weeks.

ARM II: Patients meet with therapist over 60 minutes for 2 sessions and phone calls over 15 minutes once weekly for 4 weeks.

After completion of study, patients are followed up at 1, 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed head and neck squamous cell carcinoma who have a CRT treatment scheduled at Roswell Park
* Age >= 18 years of age
* Able to read, comprehend and speak the English language
* Willing to wear a wristwatch (actiwatch) and complete the sleep log to monitor sleep and activity for three weeks (Week 1, 3, and 6) during CRT
* Willing to wear the ApneaLink Air at-home sleep monitor for one night at baseline (pre-CRT)
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* Willing to provide biospecimen samples (saliva, cheek cells, and blood) twice during CRT (week 1 and week 4) and optional for week 6
* ADDITIONAL INTERVENTIONAL STUDY CRITERIA
* Insomnia Severity Index (ISI) total score >= 7
* Willing to complete a course of Brief Behavioral Therapy for Insomnia (BBT-CI) during the treatment weeks

Exclusion Criteria:

* Participant does not meet the overall Inclusion Criteria for this study
* Patients who developed severe oral mucositis with World Health Organization Scale III or above with ulcers on the cheeks
* ADDITIONAL INTERVENTION STUDY (BBT-CI): Currently receiving treatment for insomnia or other sleep disorders
* ADDITIONAL INTERVENTION STUDY (BBT-CI): History of severe mental illness
* ADDITIONAL INTERVENTION STUDY (BBT-CI): Attending behavioral intervention programs for smoking cessation or other substance use disorders
* ADDITIONAL INTERVENTION STUDY (BBT-CI): Shift workers or persons with a known sleep disorder affecting regular sleep phase initiation (e.g. sleep onset outside the 9 pm- 12 am hours)
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the participant an unsuitable candidate for study participation
* Cognitively impaired adults/adults with impaired decision-making capacity, individuals who are not yet adults (infants, children, and teenagers), pregnant women, and prisoners are all excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Development of oral mucositis (OM) | Up to 1 year
  OM is assessed weekly during treatment by clinical exam and patient reported Oral Mucositis Weekly Questionnaire-Head and Neck Cancer (OMWQ-HN).
Self-reported oral mucositis pain | Up to 1 year
  OM pain is assessed using a visual analog scale that rates patients' overall mouth and throat soreness, on a scale of 0-10, weekly during CRT and after chemoradiotherapy (CRT) up to one year at follow up visits.
Insomnia Severity Index (ISI) | Up to 1 year
  A brief questionnaire where the total responses are added up with higher scores indicating more acute symptoms of insomnia.
Sleep Efficiency | Up to 1 year
  Will be measured by using a non-invasive wrist actigraphy monitor.
Sleep Disturbance | Up to 1 year
  Sleep diaries will assess sleep and wake time

SECONDARY OUTCOMES:
Systemic inflammatory markers will include IL-6, IL1b and TNF. | Up to 1 year
Correlation of sleep measurement with total opioid use | Up to 1 year
  Opioids are carefully prescribed as standard of care during CRT according to the severity of pain. Total opioid use, summarized by morphine milligram equivalents, will therefore also be assessed as a surrogate for overall pain severity.

CONTACTS AND LOCATIONS:
Overall Officials: Fangyi Gu, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States